CLINICAL TRIAL: NCT03135795
Title: The Influence of Epigenetic Modification in OPRM1 on Postoperative Analgesia and Side Effect Induced by μ-opioid Receptor Agonists
Brief Title: The Epigenetic Modification in OPRM1 on Postoperative Analgesia and Side Effect Induced by Sufentanil
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Ai Ling, attending doctor, Huazhong University of Science and Technology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: ALing
Record Dates: First submitted 2017-03-01; First posted 2017-05-01 (Actual); Last update posted 2017-05-01 (Actual); Status verified 2017-04

CONDITIONS: Epigenetics
Keywords: sufentanil; DNA methylation
MeSH Terms: interventions — Sufentanil; Dexmedetomidine; Propofol; Rocuronium; Sevoflurane; Remifentanil; parecoxib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- patients undergoing pancreatectomy (Experimental): patients undergoing pancreatectomy received dexmedetomidine 1μg/Kg，sufentanil 0.5μg/Kg， propofol 2mg/Kg，rocuronium 0.6mg/Kg for induction.And received sevoflurane(1-2%), remifentanil(0.1-0.2ug/kg/min) and propofol(0.3-0.6mg/kg/h) for maintenance. Parecoxib 40mg was given single intravenously before incision. And PCA with sufentanil 1ug/ml was started immediately after surgery.
  Interventions: Drug: Sufentanil; Drug: dexmedetomidine; Drug: propofol; Drug: Rocuronium; Drug: sevoflurane; Drug: remifentanil; Drug: Parecoxib

INTERVENTIONS:
Drug: Sufentanil — Patients received intravenous sufentanil 0.5μg/kg for induction,and received PCA after surgery with sufentanil 1ug/ml using a controlled infusion pump, which was programmed to use a loading dose of 2ml, background infusion at 2m/h, PCA dose of 1ml, lockout time of 10min, and maximal dose of 12ml within 1 hour period.
  Other Names: Sufentanil Citrate Injection
Drug: dexmedetomidine — Patients received intravenous dexmedetomidine 1μg/Kg for induction.
  Other Names: Dexmedetomidine Hydrochloride Injection
Drug: propofol — Patients received intravenous propofol 2mg/Kg for induction, and received intavenous pump of propofol (0.3-0.6mg/kg/h) for maintenance.
  Other Names: propofol injection
Drug: Rocuronium — Patients received intravenous rocuronium 0.6mg/Kg for induction.
  Other Names: Rocuronium Bromide Injection
Drug: sevoflurane — Patients received inhalation of sevoflurane (1-2%) for maintenance.
Drug: remifentanil — Patients received intavenous pump of remifentanil (0.1-0.2ug/kg/min) for maintenance.
  Other Names: remifentanil Citrate Injection
Drug: Parecoxib — Parecoxib 40mg was given single intravenously before incision.
  Other Names: Dynastat

SUMMARY:
To explore the epigenetic mechanism of postoperative analgesia and side effect induced by μ-opioid Receptor Agonists presented with sufentanil among general population.

DETAILED DESCRIPTION:
Patients were interviewed the day before surgery, and taught about the use of PCA pump and VAS. Pressure pain threshold(PPT) and pressure pain tolerance(PTO) were collected before surgery.

Dexmedetomidine1μg/Kg，sufentanil 0.5μg/Kg， propofol 2mg/Kg and rocuronium 0.6mg/Kg were given intravenously for induction. Anesthesia was maintained with inhalation of 1% sevoflurane and infusion of remifentanil (0.2-0.4ug/kg/min) and propofol (6-10mg/kg/h). Aterial blood pressure(ABP)，central venous pressure(CVP)，SPO2， HR，ETCO2，T and Narcotrend were monitored. Before incision, parecoxib 40mg was given intravenously, and PCA with sufentanil 1ug/ml was started immediately after surgery, suing a controlled infusion pump. The pump was programmed to use a loading dose of 2ml, background infusion at 2m/h, PCA dose of 1ml, lockout time of 10min, and maximal dose of 12ml with 1 h period.

VAS(static), VAS(dynamic), Ramssay, HR, NBP, SpO2, PCA pressing frequency, PCA comsumption were recorded 6h, 12h, 24h, 48h after surgery. Side effects such as nausea, vomiting, respiratory depression; pruritus; abdominal distention; urinary retention and dizziness were also recorded, and corresponding treatment were given.

EDTA anti-coagulated blood was collected from a central venous catheter during the operation. Genomic DNA was extracted from the blood samples, and characteristics and degree of DNA methylation of the gene OPRM1 were analysed.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical status Ⅰ-Ⅱ ;
* Weight 50-75 kg;

Exclusion Criteria:

* Long history of alcohol or analgesic drugs(including opioid ) abuse;
* Heavy smoking;
* Motion sickness;
* Long history of PONV;
* Chronic pain;
* Complicated with severe heart、brain or kidney disease.

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-02-06 (Actual); Primary Completion 2017-05-31 (Estimated); Study Completion 2017-05-31 (Estimated)

PRIMARY OUTCOMES:
Quantification of methylation in CpG islands located in gene OPRM1 | 3 months
  EDTA anti-coagulated blood was collected before induction. Genomic DNA was extracted according to the manufacturer's protocol, and CpG islands in the OPRM1 gene region were identified by CpG Island Explorer 2.0 software. Quantification of DNA methylation of all CpG sites from position +528 to +1649 in CpG islands was analysed.

SECONDARY OUTCOMES:
Pressure pain threshold (PPT) and pressure pain tolerance (PTO) | 1 day
  Patients' Pressure pain threshold(PPT) and pressure pain tolerance(PTO) in Kg/cm2 were measured before surgery using electronic pressure algometer (YISIDA-DS2, Hongkong, China).
Sex | 1 day
  Patients' sex (male or female) was recorded before surgery.
Age | 1 day
  Patients' age in years was recorded before surgery.
Weight | 1 day
  Patients' weight in kilograms was recorded before surgery.
Height | 1 day
  Patients' height in meters was recorded before surgery.
History of smoking | 1 day
  Patients' history of smoking (yes or no) was recorded before surgery.
VAS (static) and VAS (dynamic) | 6hours, 12hours, 24hours, 48hours after surgery.
  Patients' VAS(static) and VAS(dynamic) score (range 0-10) were recorded at time point of 6hours, 12hours, 24hours, 48hours after surgery.
Ramssay | 6hours, 12hours, 24hours, 48hours after surgery.
  Patients' Ramssay score (range 1-6) was recorded at time point of 6hours, 12hours, 24hours, 48hours after surgery.
Heart rate (HR) | 6hours, 12hours, 24hours, 48hours after surgery
  Patients' HR in bpm was recorded at time point of 6hours, 12hours, 24hours, 48hours after surgery.
Blood pressure (BP) | 6hours, 12hours, 24hours, 48hours after surgery.
  Patients' BP in mmHg was recorded at time point of 6hours, 12hours, 24hours, 48hours after surgery.
Pulse oxygen saturation (SpO2) | 6hours, 12hours, 24hours, 48hours after surgery.
  Patients' SpO2 in percent was recorded at time point of 6hours, 12hours, 24hours, 48hours after surgery.
PCA pressing frequency | 6hours, 12hours, 24hours, 48hours after surgery
  Patients' PCA pressing frequency in time was recorded at time point of 6hours, 12hours, 24hours, 48hours after surgery.
PCA consumption | 6hours, 12hours, 24hours, 48hours after surgery
  Patients' PCA consumption in ml was recorded at time point of 6hours, 12hours, 24hours, 48hours after surgery.
Side effects | 6hours, 12hours, 24hours, 48hours after surgery
  Side effects such as nausea, vomiting, respiratory depression, pruritus, abdominal distention, urinary retention and dizziness (yes or no) were recorded at time point of 6hours, 12hours, 24hours, 48hours after surgery, and corresponding treatment were given.

CONTACTS AND LOCATIONS:
Overall Officials: Xu Hui, Study Chair — Department of Anaesthesiology, Tongji Hospital of Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Department of Anaesthesiology, Tongji Hospital of Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No